CLINICAL TRIAL: NCT01685619
Title: A Multi-Centre Observational Prospective Cohort Study Involving the Collection of Clinical Information and Biological Specimens for the Evaluation of Novel Prognostic Tests for Myelodysplasia and Acute Myeloid Leukemia
Brief Title: AML-MDS Novel Prognostic Tests Clinical Study
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Terry Fox Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AML-MDS 01-2011
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: AML; Acute Myeloid Leukemia; MDS; Myelodysplastic Syndrome; Prognostic; Economic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Some of the laboratory tests that will be evaluated as part of this study will utilize RNA and/or DNA. There may be biospecimens left over after the work related to this study is complete. At the time of consent for the study, participants will be asked to provide consent (or decline their consent) regarding the use of leftover specimens (including RNA and DNA) for other research. The details regarding this other research are provided in the protocol and consent template.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AML Cohort: This cohort is comprised of participants who have acute myelogenous leukemia (AML).
- MDS Cohort: This cohort is comprised of participants who have myelodysplastic syndrome (MDS).

SUMMARY:
This clinical study will provide the study specimens (samples of bone marrow and blood) and the clinical data for a pan-Canadian collaborative research project developed by the MDS/AML Research Consortium. The goal of this project involves the evaluation and potential validation of five novel prognostic tests for myelodysplasia (MDS) and/or acute myeloid leukemia (AML), as well as an analysis of health economic and socio-ethical implications related to the potential introduction of these tests into the clinical setting. The over-arching goal is to improve the outcomes of patients with MDS and AML. The primary hypothesis is that one or more of the laboratory tests being evaluated in conjunction with this study, either alone or in combination with other laboratory tests (either established or under investigation in this project), will have statistically significant prognostic value either alone or in combination with established clinical risk factors.

The clinical study will involve the enrollment of 200 adults with AML and 200 adults with MDS over a 2.5 year period. Participants will be followed on study for two years. Bone marrow and blood specimens will be collected at diagnosis and at other time points as required for the development of the five laboratory tests.

Participants will be assigned to treatment according to local institutional practice and will be followed for up to 2 years. Health economic and quality of life questionnaires will be administered at key time points. Data will be collected regarding participant characteristics, diagnosis, disease features, treatment and clinical outcome.

DETAILED DESCRIPTION:
Two of the tests involve a technology called flow cytometry. Both of the flow cytometry tests are used to predict whether a person is likely to have a good response to chemotherapy or not.

Three of the tests involve new genetic-based technology. One of these tests is called comparative genomic profiling. This test can detect genetic abnormalities that current testing methods are not able to detect. Another test involves micro-RNA profiling. The final test involves RNA sequencing. The researchers think these tests might be useful in predicting how well a person will respond to treatment.

The novel laboratory tests being evaluated as part of this study are still in the early phases of development and cannot be used for clinical decision making. Participants enrolled in this study will not be informed regarding their individual results with respect to the study tests that are conducted using their biospecimens.

The following information (data) will be collected regarding study participants: diagnosis, results of relevant clinical tests, age, gender, treatment and outcome during the 2 year study follow-up period. The study also involves the completion of study questionnaires at six different time points over the course of the two year study follow-up.

ELIGIBILITY:
There are two parts to the study: Part One (Collection of Biospecimens) and Part Two (Two year follow-up that includes data collection regarding treatment, outcome and questionnaire completion).

INCLUSION CRITERIA (PART ONE):

Prospective participants can be included in the study if:

* The participant is 18 years of age or older
* The participant is suspected to have a new diagnosis of MDS (including CMML) , OR suspected to have a new diagnosis of AML excluding acute promyelocytic leukemia (APL), OR known to have a diagnosis of MDS (including CMML) confirmed by bone marrow aspirate and biopsy no more than one year prior to the date of enrollment AND without commencement of definitive therapy prior to enrollment
* The participant is scheduled to have a diagnostic or confirmatory bone marrow aspirate and biopsy at a participating site, or in the case of prospective participants with an established diagnosis of MDS (including CMML), must be able to undergo a bone marrow aspirate for the study at the participating site
* The participant must be able to read and/or understand spoken English or French so that they will be eligible for Part Two of the study
* The participant must be able to understand and sign the informed consent form applicable to their situation

EXCLUSION CRITERIA (PART ONE):

Prospective participants should be excluded from the study if:

* The participant has already received definitive therapy for AML or MDS
* The participant has a diagnosis of MDS that was confirmed more than one year prior to the date of enrollment

INCLUSION CRITERIA (PART TWO):

Participants who have been enrolled in Part One will be eligible to participate in the full two year study follow-up component if they meet the following criteria:

* Confirmed diagnosis of either MDS, CMML or AML (excluding APL)
* Sufficient cell count for the MDS/AML Clinical Study requirements as follows:

For participants with suspected (or known) AML:

The blast count of the peripheral blood taken at diagnosis must be greater than 1 x10^6 blast count/mL

* It must be possible to earmark for the MDS/AML Study:
* 3 vials 1.0 x 10^7/mL mononuclear peripheral blood cells
* 1 vial 0.5 x 10^7/mL mononuclear bone marrow cells

Cells are to be prepared according to the site's local cell bank procedures so that they can be stored and transported to study labs as needed.

At sites participating in the Hogge Assay:

In addition to the specimens described above, it must be possible to provide 2 mL of fresh bone marrow or 5 mL of fresh peripheral blood with > 1 x 10^6 blast count/mL

For participants with suspected (or known) MDS:

* It must be possible to earmark for the MDS/AML Study:
* 2 vials 1.0 x 10^7/mL mononuclear peripheral blood cells
* 2 vials 1.0 x 10^7/mL mononuclear bone marrow cells

Cells are to be prepared according to the site's local cell bank procedures so that they can be stored and transported to study labs as needed.

EXCLUSION CRITERIA (PART TWO):

Participants who have been enrolled in Part One will not be eligible to participate in the full two year study follow-up component if they:

* Do not have sufficient cell count for the MDS/AML Clinical Study requirements as set out in Section 11.3
* It is confirmed after enrollment that they do not have a diagnosis of MDS, CMML or AML
* A diagnosis of APL is confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective participants will include patients with known or supsected AML or MDS who are being treated and/or assessed at a participating site.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-10-02 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Prognostic capacity of the candidate tests (alone and in combination) to predict response to treatment, time to relapse, time to death. | Two years following the completion of enrollment.
  For the AML cohort, the candidate prognostic tests will be analyzed with adjustments for following clinical factors: age, white blood cell count at presentation, antecedent hematologic disorder, FLT-3 status, Karnofsky Performance Status (KPS), cytogenetic sub-group (using WHO 2008). For the MDS cohort the candidate prognostic tests will be analyzed with adjustments for following clinical factors: age, KPS, karyotype, bone marrow blast count and number of cytopenias at diagnosis.

SECONDARY OUTCOMES:
Cost impact of candidate tests. | Two years following the completion of enrollment.
  The cost-effectiveness of the candidate tests for AML and MDS treatment will be projected with the aid of economic simulation models.
Societal risks and benefits related to the candidate tests. | Two years following the completion of enrollment.
  A comparative analysis of policies and regulations in Canada governing prognostic tests will be undertaken (including tests that utilize RNA and DNA based technologies). In addition, input will be obtained from key stakeholders. This information will be used to develop a set of guidelines and best practices for this type of research.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Couban, M.D., Principal Investigator — Nova Scotia Health Authority
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre (formerly Princess Margaret Hospital), Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec